CLINICAL TRIAL: NCT07390565
Title: Yishen Qutong Granules Combined With Immunochemotherapy for Extensive-Stage Small Cell Lung Cancer: A Multicentre, Randomised, Triple-Blind, Placebo-Controlled Trial
Brief Title: YSQTG Combined With Immuno-chemotherapy for Extensive-Stage Small Cell Lung Cancer
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: LI FENG (Other)
Collaborators: Henan Cancer Hospital (Other Government); Fudan University (Other); Shanxi Province Cancer Hospital (Other)
Responsible Party: Sponsor-Investigator, LI FENG, Consultant Physician, Professor, Doctoral Supervisor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Organization: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025YFC3508301
Record Dates: First submitted 2026-01-22; First posted 2026-02-05 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-07

CONDITIONS: Extensive-stage Small Cell Lung Cancer (SCLC)
Keywords: Traditional Chinese Medicine; Western Medicine
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group(Yishen Qutong Granules) (Experimental): Yishen Qutong Granules administered at 10g per dose, three times daily, in conjunction with immunotherapy plus etoposide and platinum-based first-line treatment.
  Interventions: Drug: Yishen Qutong Granules
- Control group(Placebo) (Experimental): In parallel with immunotherapy plus etoposide and platinum-based first-line treatment, administer a simulated formulation of Yishen Qutong Granules (1/10 Yishen Qutong Granules), 10g per dose, three times daily.
  Interventions: Drug: Yishen Qutong Simulant Granules

INTERVENTIONS:
Drug: Yishen Qutong Granules — The patent prescription of Professor Feng Li, the head of the Department of Traditional Chinese Medicine at the Cancer Hospital of the Chinese Academy of Medical Sciences.
  Arms: Treatment group(Yishen Qutong Granules)
Drug: Yishen Qutong Simulant Granules — Yishen Qutong Simulant Granules is a preparation with one-tenth the dosage of Yishen Qutong Granules.
  Arms: Control group(Placebo)

SUMMARY:
Globally, lung cancer stands as the foremost cause of cancer-related mortality. Among its subtypes, small cell lung cancer (SCLC) represents an exceptionally aggressive malignancy, accounting for approximately 15-20% of all lung cancer cases. Over two-thirds of SCLC patients are diagnosed at an extensive stage, facing a median survival of only 7-12 months, a 2-year survival rate below 5%, and a dismal 5-year survival rate of 2%, underscoring its poor prognosis and high mortality. First-line treatment for extensive-stage SCLC typically involves comprehensive therapy centered on chemotherapy, often combined with immunotherapy. While this approach can achieve response rates of 50-70%, it is frequently accompanied by significant adverse effects, including bone marrow suppression and debilitating gastrointestinal reactions such as nausea, vomiting, and anorexia. The considerable toxicity associated with chemotherapy poses a major clinical challenge, limiting the potential for dose or duration escalation and hindering further efficacy gains. Therefore, developing strategies to mitigate toxicity while enhancing therapeutic efficacy remains an urgent clinical priority.

In the paradigm of Traditional Chinese Medicine (TCM), extensive-stage SCLC is categorized under syndromes such as "pulmonary accumulation," "cough," and "consumptive disease." Its fundamental pathogenesis is characterized by a deficiency of healthy qi (vital energy) alongside an excess of pathogenic factors, primarily "toxins," "stasis," and "phlegm." The core pathological mechanism involves the internal accumulation of toxins, disruption of the lung's dispersing and descending functions, disharmony of qi and blood, and consequent depletion of vital qi over time. Treatment strategies thus aim to resolve toxins, dispel stasis, and reinforce the body's vital qi. Preliminary clinical observations suggest that the TCM formula Yishen Qutong Granules, developed based on the theories of "reinforcing healthy qi to resolve toxins" and the "metal-water mutual generation" principle, can significantly alleviate symptoms in SCLC patients. Building on this foundation, the present study proposes to evaluate the integration of Yishen Qutong Granules with standard chemo-immunotherapy for extensive-stage SCLC, with the objectives of improving patients' quality of life and extending overall survival.

To this end, investigators will conduct a multicenter, randomized, triple-blind, placebo-controlled clinical trial. A total of 308 patients with extensive-stage SCLC, who are scheduled to undergo first-line immunotherapy combined with etoposide and platinum-based chemotherapy, will be enrolled from participating centers. Participants will be randomly allocated in a 1:1 ratio to either the treatment group or the control group (n=154 each). The treatment group will receive oral Yishen Qutong Granules (10g, three times daily) in addition to the standard chemo-immunotherapy regimen. The control group will receive an identical regimen of standard therapy along with a matched placebo granule. The intervention period for the herbal preparation/placebo is 90 days, and all patients will be followed for 18 months. The primary efficacy endpoint is the Disease Control Rate (DCR). Secondary endpoints include Overall Survival (OS), Progression-Free Survival (PFS), TCM syndrome score (assessed using a validated scale), St. George's Respiratory Questionnaire (SGRQ) score, EORTC QLQ-C30 quality of life score, cancer-related fatigue, and emotional status. Safety will be rigorously monitored through serial assessments of routine blood/urine/stool tests, hepatic and renal function panels, and electrocardiograms. This study aims to generate high-level evidence for the integrative TCM-Western medicine approach and elucidate the potential role of Yishen Qutong Granules in the comprehensive management of extensive-stage SCLC.

ELIGIBILITY:
Inclusion Criteria:

* Meets Western medical diagnostic criteria for extensive-stage small cell lung cancer and Chinese medicine diagnostic criteria for kidney deficiency with qi deficiency and stagnation of blood stasis;
* Newly diagnosed extensive-stage small cell lung cancer patients who have not previously received Western medical antineoplastic therapy, with evaluable lesions;
* Intended to receive ≥2 cycles of first-line immunotherapy plus platinum-based chemotherapy plus etoposide;
* No concurrent or prior history of other primary malignancies;
* Aged ≥18 years with an estimated survival period of ≥3 months;
* Karnofsky Performance Status (KPS) ≥60 points;
* Normal cognitive function sufficient to complete questionnaires;
* Voluntary acceptance of the study treatment regimen and signing of informed consent.

Exclusion Criteria:

* Pregnant or breastfeeding women, or individuals with severe diseases affecting the cardiovascular, pulmonary, hepatic, renal, or haematological systems;
* Participants in other clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Estimated)
Dates: Start 2026-02-17 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Disease Control Rate（DCR） | Follow-up visits were conducted at 43 days, 90 days, 133 days, 233 days, 365 days (12 months), 450 days (15 months), and 540 days (18 months) after commencement, totalling seven visits.
  Disease Control Rate (DCR) = (Complete Response + Partial Response + Stable Disease) /Total Number of Patients × 100%

SECONDARY OUTCOMES:
Overall Survival（OS） | Before treatment commencement; 21 days after commencement; 43 days after; 90 days after; 133 days after; 233 days after; 365 days after; 450 days after; 540 days after
  The period from the commencement of treatment until the patient's death from any cause
progression-free survival（PFS） | Before treatment commencement; 21 days after commencement; 43 days after; 90 days after; 133 days after; 233 days after; 365 days after; 450 days after; 540 days after
  Time from study entry to first radiographic evidence of tumour progression
Evaluation of Syndrome and Symptom Points of Traditional Chinese Medicine | Before treatment commencement, and at 21 days, 43 days, and 90 days after commencement
  The TCM Syndrome Score evaluates the severity of symptoms related to nodule accumulation, localized pain, tongue appearance, lumbar debility, and fatigue. Each symptom is scored from 0 to 6, with higher scores indicating more severe symptoms. The total score is the sum of individual symptom scores, reflecting the overall severity of TCM syndromes.
Quality of Life assessed by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) | Before treatment commencement, and at 21 days, 43 days, and 90 days after commencement
  The EORTC QLQ-C30 is a 30-item questionnaire evaluating cancer patients' quality of life across multiple dimensions, including physical, emotional, cognitive, and social functioning, as well as symptom burden (e.g., fatigue, pain, nausea). Scores range from 0 to 100, with higher scores in functional scales and global health status indicating better quality of life, and higher scores in symptom scales indicating worse symptoms.
St George' s Respiratory Questionnaire (SGRQ) | Before treatment commencement, and at 21 days, 43 days, and 90 days after commencement
  The St George's Respiratory Questionnaire (SGRQ) is a standardised self-assessment tool used to evaluate the quality of life in patients with chronic respiratory diseases. By quantifying the impairment experienced by patients in terms of symptoms, functional capacity, and psychosocial adjustment, it comprehensively reflects the impact of the disease on patients' daily lives.
  Scale Range and Interpretation Total score range: 0 to 100. Higher scores indicate greater impairment of health-related quality of life due to respiratory symptoms.
Fatigue-Related Quality of Life (FACIT-F scale) | Before treatment commencement, and at 21 days, 43 days, and 90 days after commencement
  Cancer-related fatigue was assessed using the Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) scale.
  Scale Range and Interpretation Total score range: 0 to 52. Higher scores indicate better fatigue-related quality of life (i.e., less fatigue and its impact).
Brief Fatigue Inventory scale (BFI scale) | Before treatment commencement, and at 21 days, 43 days, and 90 days after commencement
  Fatigue severity was assessed using the Brief Fatigue Inventory (BFI) scale. Scale Range and Interpretation Total score range: 0 to 10. Higher scores indicate more severe fatigue.
Anxiety subscale of the Hospital Anxiety and Depression Scale (HADS-A) | Before treatment commencement, and at 21 days, 43 days, and 90 days after commencement
  Anxiety was assessed using the Anxiety subscale of the Hospital Anxiety and Depression Scale (HADS-A).
  Scale Range and Interpretation Total score range: 0 to 21. Higher scores indicate more severe anxiety symptoms.
Depression subscale of the Hospital Anxiety and Depression Scale (HADS-D) | Before treatment commencement, and at 21 days, 43 days, and 90 days after commencement
  Depression was assessed using the Depression subscale of the Hospital Anxiety and Depression Scale (HADS-D).
  Scale Range and Interpretation Total score range: 0 to 21. Higher scores indicate more severe depressive symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences/Peking Union Medical College, Beijing, Chaoyang, China

IPD SHARING:
Plan to Share IPD: No
The project involves some patents that will not be disclosed at this time.

REFERENCES:
- [Result] Qin K, Gay CM, Byers LA, Zhang J. The current and emerging immunotherapy paradigm in small-cell lung cancer. Nat Cancer. 2025 Jun;6(6):954-966. doi: 10.1038/s43018-025-00992-5. Epub 2025 Jun 5. PMID 40473974
- [Result] Xie M, Vuko M, Rodriguez-Canales J, Zimmermann J, Schick M, O'Brien C, Paz-Ares L, Goldman JW, Garassino MC, Gay CM, Heymach JV, Jiang H, Barrett JC, Stewart RA, Lai Z, Byers LA, Rudin CM, Shrestha Y. Molecular classification and biomarkers of outcome with immunotherapy in extensive-stage small-cell lung cancer: analyses of the CASPIAN phase 3 study. Mol Cancer. 2024 May 30;23(1):115. doi: 10.1186/s12943-024-02014-x. PMID 38811992
- [Result] Shields MD, Chiang AC, Byers LA. Top advances of the year: Small cell lung cancer. Cancer. 2025 Mar 15;131(6):e35770. doi: 10.1002/cncr.35770. PMID 40040254
- [Result] Zugazagoitia J, Paz-Ares L. Extensive-Stage Small-Cell Lung Cancer: First-Line and Second-Line Treatment Options. J Clin Oncol. 2022 Feb 20;40(6):671-680. doi: 10.1200/JCO.21.01881. Epub 2022 Jan 5. PMID 34985925
- [Result] Chen Y, Li H, Fan Y. Shaping the tumor immune microenvironment of SCLC: Mechanisms, and opportunities for immunotherapy. Cancer Treat Rev. 2023 Nov;120:102606. doi: 10.1016/j.ctrv.2023.102606. Epub 2023 Aug 7. PMID 37579532
- [Result] Zhu L, Qin J. Predictive biomarkers for immunotherapy response in extensive-stage SCLC. J Cancer Res Clin Oncol. 2024 Jan 20;150(1):22. doi: 10.1007/s00432-023-05544-x. PMID 38245636
- [Result] Tomic K, Vranic S. Small cell lung cancer (SCLC): At the door of targeted therapies. Biomol Biomed. 2025 Aug 29;26(1):1-4. doi: 10.17305/bb.2025.13195. PMID 40884462
- [Result] Kim SY, Park HS, Chiang AC. Small Cell Lung Cancer: A Review. JAMA. 2025 Jun 3;333(21):1906-1917. doi: 10.1001/jama.2025.0560. PMID 40163214